CLINICAL TRIAL: NCT05441774
Title: Stimulating Compassion: Using Transcutaneous Vagus Nerve Stimulation (tVNS)
Brief Title: Stimulating Compassion UsingTranscutaneous Vagus Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 07760/006
Record Dates: First submitted 2022-06-23; First posted 2022-07-01 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers
Keywords: Vagus nerve; Neurostimulation; Transcutaneous vagus nerve stimulation; Mental imagery; Compassion; Meditation

STUDY DESIGN:
Intervention Model Description: Factorial 2 (sham stimulation v active stimulation) x 2 (sham v self-compassion imagery)
Who Masked: Participant
Masking Description: Study design and aims will be concealed from participants. They will not be made aware of the presence of active versus sham conditions (all participants are given the expectation of active stimulation and imagery).
  Participants are informed of their imagery condition before consent is obtained on the first lab session.
  Study aims will be disclosed at debriefing, after all experimental procedures have been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sham stimulation plus sham imagery (Sham Comparator): Double sham group: Stimulator electrodes will be applied to earlobe (sham stimulation); imagery task will involve a 'draw-a-face-in-imagination' (sham imagery) task.
  Interventions: Device: Sham transcutaneous vagus nerve stimulation; Behavioral: Sham mental imagery
- Active stimulation plus sham imagery (Other): Single (imagery) sham group: Stimulator electrodes will be applied to the tragus (active stimulation); 'draw-a-face-in-imagination' (sham imagery) task.
  Interventions: Device: Active transcutaneous vagus nerve stimulation; Behavioral: Sham mental imagery
- Sham stimulation plus active self-compassion imagery (Other): Single (stimulation) sham group: earlobe (sham) stimulation; imagery task will involve directing compassion to the self (self-compassion, active imagery).
  Interventions: Behavioral: Active self-compassion imagery; Device: Sham transcutaneous vagus nerve stimulation
- Active stimulation plus active self-compassion imagery (Active Comparator): Double active group: tragus (active) stimulation; self-compassion (active imagery)
  Interventions: Device: Active transcutaneous vagus nerve stimulation; Behavioral: Active self-compassion imagery

INTERVENTIONS:
Device: Active transcutaneous vagus nerve stimulation — TVNS is a non-invasive counterpart to surgical methods for stimulating the vagus. For the active condition, stimulator electrodes deliver a mild electrical current to the tragus. Stimulation parameters: stimulation of left tragus via two gold-plated electrodes, attached by ear-clip. Waveform: rectangular, frequency: 20 Hz, pulse width: 0.2 ms, individually adjusted intensity based on participant's perceptual threshold.
  Other Names: Parasym tVNS device
  Arms: Active stimulation plus active self-compassion imagery; Active stimulation plus sham imagery
Behavioral: Active self-compassion imagery — Self-compassion imagery is both a meditative technique and a component of compassion-focused cognitive therapy. Here, self-compassionate imagery is delivered as standardized audio-recorded instructions.
  Arms: Active stimulation plus active self-compassion imagery; Sham stimulation plus active self-compassion imagery
Device: Sham transcutaneous vagus nerve stimulation — TVNS is a non-invasive counterpart to surgical methods for stimulating the vagus. For the sham condition, stimulator electrodes deliver a mild electrical current to the earlobe. Stimulation parameters: stimulation of left earlobe via two gold-plated electrodes, attached by ear-clip. Waveform: rectangular, frequency: 20 Hz, pulse width: 0.2 ms, individually adjusted intensity based on participant's perceptual threshold.
  Other Names: Parasym tVNS device
  Arms: Sham stimulation plus active self-compassion imagery; Sham stimulation plus sham imagery
Behavioral: Sham mental imagery — Draw-a-face-in-imagination is the sham/ control imagery condition. Here, control imagery instructions are delivered as a standardized audio-recording, well-matched to self-compassion imagery for number of words, complexity of language, and duration of the audio instructions.
  Arms: Active stimulation plus sham imagery; Sham stimulation plus sham imagery

SUMMARY:
This experimental proof-of-concept study in healthy volunteers investigates whether a specific form of self-relating, namely, self-compassion, can be controlled through non-invasive stimulation of the vagus nerve. The vagus nerve is part of the parasympathetic nervous system (the 'rest and digest' system) and its fibers are spread throughout the upper body, face, and neck, including a branch that innervates parts of the external ear (e.g. the tragus), close to the surface of the skin. This allows the 'auricular branch' of the vagus nerve to be readily stimulated electrically. Importantly, this can be achieved non-invasively using a transcutaneous vagus nerve stimulation (tVNS) device. The investigators will test the effects of tVNS alone and in combination with a meditation-like technique that is intended to increase participants' feelings of self-compassion (self-compassion imagery). In particular, the investigators will assess participants' experience of self-compassion and self-criticism, as well as other outcome measures, before and during stimulation, and again after they perform the self-compassionate imagery exercise. These effects will be compared to three other groups: one that receives tVNS along with a control (sham) imagery procedure, another that receives sham tVNS and self-compassion imagery, and a final group that receives sham tVNS and sham imagery. It is expected that the group that receives active tVNS and the self-compassion imagery exercise will experience the largest average increases in self-compassion and decreases in self-criticism. The findings of this study will help us better understand the role of the vagus nerve in complex cognitive-emotional experiences - like compassion - and may also motivate the development of bioelectronic stimulation methods that can be used alongside psychological techniques for improving self-compassion and reducing self-criticism, particularly among people with certain psychological disorders.

DETAILED DESCRIPTION:
The role of the vagus nerve in regulating cardiac, respiratory, and gut functioning via brainstem nuclei is well-established. More recently, its role has been examined in relation to the modulation of higher cognitive functions. Bodily signals (e.g. from the heart or gut) conveyed by vagal afferents could affect cognitive functioning via projections from the nucleus of the solitary tract (NTS) to the locus coeruleus and thence to widespread cortical areas through noradrenergic outputs. In addition, the NTS transmits sensory-visceral information to the central autonomic network, which includes higher brain areas (e.g. prefrontal cortex). Recent research suggests that vagus nerve activity is associated with a range of psychological functions including memory, executive function, and threat/fear processing. In addition, biobehavioral theories of vagal functioning, and emerging empirical evidence suggest a role for the vagus nerve in modulating social behavior as well as complex emotional states.

A number of researchers have proposed a role for vagal nerve functioning in well-being, and particularly in generating or modulating feelings of 'safeness', contentedness, and relaxation that underlie complex social-affective-motivational states, such as compassion. Previous research has examined the effects of inducing compassionate feelings while measuring vagus nerve activity (via heart rate variability). However, to our knowledge, no published study has demonstrated an association between vagal activity and compassion by directly modulating the vagus nerve itself. Such studies have important theoretical implications but are also potentially valuable in the future development of interventions that employ tVNS or similar technology to augment psychological treatments that employ compassion-focused techniques (e.g. compassionate mind training; compassion-focused cognitive therapy; loving-kindness meditation-based treatments, etc.)

The current experiment aims to determine if vagus nerve activation using tVNS is sufficient to generate positive affective states, especially compassion (specifically, self-reported self-compassion). Alternatively, tVNS may produce a permissive physiological context that facilitates compassionate responding. For example, tVNS may synergize the effects of a compassion-inducing behavioral intervention. To examine these possibilities, the investigators will test the separate and combined (interacting) effects of tVNS and a compassion-induction procedure (self-compassion mental imagery) compared to sham conditions, in a four-group factorial (2 x 2) design. Participants will be randomly assigned to (i) active tVNS + sham imagery, (ii) active tVNS + active self-compassion imagery, (iii) sham-tVNS + active self-compassion and (iv) sham-tVNS + sham imagery.

In addition to examining the effects of stimulation and imagery conditions on self-compassion, the investigators will also test their effects on other types of positive affect, as well as self-criticism, which is an opposing form of self-representation to self-compassion. Self-criticism is a transdiagnostic psychological marker of psychopathology, and measures of self-criticism are sensitive to the effects of compassion-focused interventions , including brief self-compassion imagery, as will be used here. Vagal activity will be indexed using heart rate variability, and effects of stimulation and imagery will additionally be tested on attentional bias (e.g. first fixation, increased dwell time) to compassionate facial expressions.

Participants attend two lab sessions (on Day 1 and 8) in which they will undergo either supervised active or sham tVNS and either the self-compassion or sham imagery exercise (delivered as standardized audio instructions), per their randomized condition. Assessments of heart rate variability, self-compassion, self-criticism, positive state affect, and state mindfulness will occur before stimulation, during stimulation, and after the imagery exercise. In addition, participants will complete the Day 1 stimulation procedure and imagery task on Days 2-7, guided via online audio and written instructions. This will allow us to test the effects of extended (daily) stimulation and imagery practice. Additional study details are available on the Open Science Framework (osf.io/k2dje).

ELIGIBILITY:
Inclusion Criteria:

* Fluency in English
* Good (including corrected) vision and hearing.

Exclusion Criteria:

* Current use of any medication for a psychiatric condition
* Regular use of any medication used to treat a cardiovascular condition or inflammation
* Use of any illicit recreational drug >2/week
* Regularly consuming >14 standard UK 'units' of alcohol
* Currently receiving treatment for any mental health condition
* Scores on screening measures of depression (PHQ-2) and/or anxiety (GAD-2) that indicate significant levels of current/recent anxiety or depression (scores on either >4)
* History of serious mental health problems (schizophrenia, bipolar disorder)
* Past or current cardiovascular or neurological problems
* Current/past problems related to chronic/recurring facial or ear pain
* Skin irritation/ broken skin at stimulation site
* Pregnancy or likelihood of becoming pregnant during study
* Previous adverse response to meditation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
State self-compassion | 1 week
  Self-compassion subscale of the scenario-based self-compassion and self-criticism Scales (SCCS; Falconer et al, 2015). Score range: 15 (minimum) to 105 (maximum). High scores indicate greater self-compassion (desirable outcome)
Heart rate variability | 1 week
  Root mean square of successive differences (commonly, RMSSD) between normal beats; high-frequency power. Higher levels indicate greater heart rate variability (a desirable outcome)
State self-criticism | 1 week
  Self-criticism subscale of the SCCS (Falconer et al, 2015). Score range: 15 (minimum) to 105 (maximum). High scores indicate greater self-criticism (undesirable outcome)

SECONDARY OUTCOMES:
Eye-tracking attention metrics | 1 week
  Dwell time, first fixation and pupillometric indices of attentional bias to compassionate facial expressions (stimuli from Falconer et al., 2019). Faces differ in intensity (25%, 50%, 75%, 100% compassion) versus matched neutral expression.
State mindfulness | 1 week
  5 items (2 body, 2 mind, and 1 activity-related mindfulness items) from the State Mindfulness Scale (Tanay & Bernstein, 2013) as used by Shohan et al (2017). The range (average across items) is 1 to 5, with high levels indicating greater state mindfulness (desirable outcome).
State positive and negative affect | 1 week
  Positive affects subscale of the International positive and negative affect schedule-SF (iPANAS, 10 item version; Thompson, 2007). Range of scores 5 (minimum) - 25 (maximum) for positive affect and 5-25 for negative affect, with higher scores indicating greater amounts of positive (desirable) and negative (undesirable) affect respectively.
State positive affect (Safe/content) | 1 week
  Safe/content positive affect subscale of the Types of Positive Affect Scale (TPAS; Gilbert et al., 2008). Range of scores: 0 (minimum) -16 (maximum), with higher levels indicating greater levels of 'safeness'/contentedness (desirable outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Sunjeev K Kamboj, PhD, Principal Investigator — UCL
Locations (1):
- Clinical Psychopharmacology Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request to PI

REFERENCES:
- [Derived] Kamboj SK, Peniket M, Simeonov L. A bioelectronic route to compassion: Rationale and study protocol for combining transcutaneous vagus nerve stimulation (tVNS) with compassionate mental imagery. PLoS One. 2023 Mar 13;18(3):e0282861. doi: 10.1371/journal.pone.0282861. eCollection 2023. PMID 36913378